CLINICAL TRIAL: NCT01738399
Title: Influence of Coffee Consumption on Insulin Sensitivity in Overweight and Insulin Resistant Subjects.
Brief Title: Coffee and Metabolic Health Outcomes
Acronym: COMETH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11.09.NRC
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2012-03

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance; Coffee; Glucose metabolism
MeSH Terms: conditions — Insulin Resistance | interventions — Coffee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coffee (Experimental): Subjects take 4 cups of coffee mix per day for 24 weeks
  Interventions: Dietary Supplement: Coffee
- Placebo (Placebo Comparator): Subjects take 4 cups of placebo per day for 24 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coffee
  Arms: Coffee
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate the long-term (24 weeks) effects of coffee consumption on insulin sensitivity in insulin resistant individuals.

DETAILED DESCRIPTION:
Coffee is a major source of the phenolic acid chlorogenic acid and a substantial source of trigonelline, niacin, lignans magnesium, and potassium. Several of these compounds have been shown to improve glucose metabolism in animal models. Consumption of coffee was inversely associated with the risk of type-2 diabetes in prospective cohort studies across the world. Consumption of 3 to 4 cups of coffee per day was associated with an approximately 25% lower risk of type-2 diabetes. However, direct evidence of the efficacy of coffee to reduce blood glucose and insulin resistance parameters in humans from randomized trials is still lacking. In recent small trials of short duration (up to 6 weeks) coffee consumption increased levels of the insulin-sensitizing hormone adiponectin, but did not significantly improve insulin sensitivity These results suggest that a larger longer-term trial of the effects of coffee consumption on directly measured insulin sensitivity is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects classified as being insulin-resistant in the screening visit. Subjects should have a non-diabetic fasting plasma glucose concentration (< 7.0 mM) and a HOMA-IR > 2.2. The HOMA-IR was demonstrated as a reliable indicator of insulin resistance strongly correlated with values obtained by clamp (4). The cut-off value of the HOMA-IR was defined according to data obtained in the Singapore cohort. It corresponds to the 75th percentile of the population. The HOMA-IR cut-off was subsequently revised to ≥ 1.3 to increase recruitment rates.
* Age: ≥ 35 to ≤ 69 years old
* Body mass index : ≥ 22.5 to ≤ 35.4 kg/m2
* Users of at least 1 cups of caffeinated coffee per day who are willing to be randomized to any of the interventions.
* Subjects should be willing to stop consuming caffeinated soft drinks or supplements during the study and to drink coffee with non-dairy creamer.
* Non-smokers (< 1 cigarette per week)
* Participants have been weight stable for at least -8 weeks pre-ceding the screening visit (± 2.5 kgs).
* Chinese, Malay and Indian ethnicity

Exclusion Criteria:

Subjects representing one or more of the following criteria are excluded from participation in the study:

* Any condition/illness that may affect the study outcomes or would make participation potentially harmful such as pregnancy or breastfeeding, diabetes mellitus, heart disease, stroke, hypertension, malabsorption syndromes, GERD, a history of ulcer, clotting or bleeding disorders,allergy to the test beverage, allergy to insulin, according to a detailed medical history.
* Participants who are allergic to foods may be excluded based on the investigator's discretion.
* Participants consume > 2 alcoholic servings/day on a regular basis and > 8 caffeinated servings (based on tea and coffee)/day
* Present drug abuse or use of medications that could interfere with the treatment including bronchodilators, quinolone antibiotics, monoamine oxidase inhibitors, anxiolytics, ranitidine, corticosteroids, growth hormone, anti-hypertensives. These conditions will be screened based on subject reporting. Participants will be asked to bring in their current medications at the time of screening, and these will be checked by the study-staff.
* Subject is taking traditional medications, herbal or dietary supplements that may affect the study outcome in the opinion of the investigators.
* Subject who cannot be expected to comply with the study procedures in the opinion of the investigators.
* Currently participating or having participated in another clinical trial during the last 12 weeks prior to the beginning of this study.
* Premenopausal women with self-reported irregular menstrual cycles or peri-menopausal women (participants who stopped getting their menses for less than 48 weeks ).

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity when compared to baseline as measured using the euglycemic hyperinsulinemic clamp. | Baseline and 24 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose concentration from baseline to 12 weeks | Baseline, 12 weeks
Change in fasting plasma glucose concentration from baseline to 24 weeks | Baseline, 24 weeks
Change in fasting plasma total adiponectin concentrations from baseline to 12 weeks | Baseline, 12 weeks
Change in fasting plasma total adiponectin concentrations from baseline to 24 weeks | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rob M van Dam, Principal Investigator — Saw Swee Hock School of Public Health, National University of Singapore
Locations (2):
- Singapore (2):
  - Saw Swee Hock School of Public Health, Singapore, Singapore
  - Saw Swee Hock School of Public Health, Singapore

REFERENCES:
- [Derived] Alperet DJ, Rebello SA, Khoo EY, Tay Z, Seah SS, Tai BC, Tai ES, Emady-Azar S, Chou CJ, Darimont C, van Dam RM. The effect of coffee consumption on insulin sensitivity and other biological risk factors for type 2 diabetes: a randomized placebo-controlled trial. Am J Clin Nutr. 2020 Feb 1;111(2):448-458. doi: 10.1093/ajcn/nqz306. PMID 31891374
- [Derived] Alperet DJ, Rebello SA, Khoo EY, Tay Z, Seah SS, Tai BC, Emady-Azar S, Chou CJ, Darimont C, van Dam RM. A randomized placebo-controlled trial of the effect of coffee consumption on insulin sensitivity: Design and baseline characteristics of the Coffee for METabolic Health (COMETH) study. Contemp Clin Trials Commun. 2016 Aug 2;4:105-117. doi: 10.1016/j.conctc.2016.06.013. eCollection 2016 Dec 15. PMID 29736473